CLINICAL TRIAL: NCT03210350
Title: Effect of Magnesium Sulphate on the Intracranial Pressure of Preeclamptic Patients Using Ultrasound Measured Optic Nerve Sheath Diameter: a Pilot Study
Brief Title: Effect of Magnesium Sulphate on the Intracranial Pressure of Preeclamptic Patients
Status: Completed | Type: Observational
Sponsor: Corniche Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CH29011702
Record Dates: First submitted 2017-06-20; First posted 2017-07-06 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2018-11

CONDITIONS: Preeclampsia Severe

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath diameter — Optic nerve sheath diameter measurement using ultrasound

SUMMARY:
It had been shown that high percentage of severe preeclampsia patients got a high cerebral perfusion pressure (CPP) due to abnormal autoregulation of cerebral blood vessels with associated endothelial dysfunction and disrupted blood brain barrier. Moreover, patients with high CPP is more likely to present with headache compared to other patients with normal CPP.In this particular scenario, use of magnesium sulphate is associated with marked reduction of CPP and. hence prevention of cerebral damage.This hypothesis was confirmed by new magnetic resonance techniques that demonstrated brain edema in eclampsia/ severe preeclampsia patient mostly due to vasogenic edema and less commonly attributed to cytotoxic edema.

Changes in the optic nerve sheath diameter (ONSD) mirrors the changes in the Intracranial pressure(ICP), subsequently when the intracranial pressure increases the optic nerve sheath diameter (ONDS) also increases.

The aim of this study is to determine the effect Magnesium sulphate infusion on intracranial pressure, in patients presented with severe preeclampsia by measuring changes in the ONSD using ultrasound examination.

DETAILED DESCRIPTION:
30 obstetric patients admitted to the HDU in Corniche Hospital for treatment of severe preeclampsia. Patients with the following criteria will be excluded from the current work: Patients undergone cranial or eye surgeries, Patients with known intracranial pathology, Patients suffering from glaucoma or any other eye pathology that prevent clear identification of the optic nerve, and Patients on drugs that may affect the cerebrospinal fluid [based on operator decision].

In this prospective pilot study, patients who will fulfill the inclusion criteria will be recruited at the time of admission in HDU by the investigators. The ONDS will be measured before the commencement of Magnesium sulphate infusion, 1hr after finishing the loading dose, 6 and 24 hrs after infusion started. Patients will be in supine position with the head of the bed less than 20 degrees. High frequency (7.5 MHz) linear probe will be used; it will be placed gently over both closed eye after liberal application of sterile gel, the patient will be instructed to look forward to align the optic nerve directly opposite to the probe. The ONSD will be measured 3mm behind the optic disc in both the sagittal and transverse planes and an average will be calculated and recorded. In the absence of complete visualization of the optic disc, the largest viewed diameter will be taken as the maximal ONSD. Hemodynamic variables & oxygen saturation will be recorded at the same times.

ELIGIBILITY:
Inclusion Criteria:

* obstetric patients admitted to the HDU at Corniche Hospital for treatment of severe preeclampsia

Exclusion Criteria:

* (1) Patients undergone cranial or eye surgeries, (2) Patients with known intracranial pathology, (3) Patients suffering from glaucoma or any other eye pathology that prevent clear identification of the optic nerve, (4) Patients on drugs that may affect the cerebrospinal fluid

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: obstetric patients admitted to the HDU at Corniche Hospital for treatment of severe preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Optic nerve sheath diameter from baseline after magnesium Sulfate administration | 1,6 and 24 hours
  Change in Optic nerve sheath diameter from baseline at 1, 6 and 24 hours after completion of Magnesium sulfate loading dose

CONTACTS AND LOCATIONS:
Locations (1):
- Corniche Hospital, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No